CLINICAL TRIAL: NCT01164956
Title: Methylphenidate for Cancer-Related Fatigue: A Pilot N-of-1 Study
Brief Title: Methylphenidate for Cancer-Related Fatigue
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient Resources
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Christina K. Ullrich, MD, MPH, Christina Ullrich, MD, MPH, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 10-146
Record Dates: First submitted 2010-07-06; First posted 2010-07-19 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Cancer
Keywords: methylphenidate; fatigue
MeSH Terms: conditions — Neoplasms; Fatigue | interventions — Methylphenidate; 5,10-dihydro-5-methylphenazine

STUDY DESIGN:
Intervention Model Description: The N-of-1 design randomized participants to 3 potential treatment pairs; Each pair incorporated the 2 drugs under investigation but with different sequence: Methylphenidate then Placebo or Placebo then Methylphenidate. With this design, there are 8 potential permutations/arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- M-P, P-M, M-P (Experimental): Participants were randomized to receive 3 treatment pairs of placebo (P) then methylphenidate (M) or M then P. Each M or P was given daily for 3 days and therefore treatment duration was 18 days over 3 treatment pairs. M or P was administered orally at a starting dose of 0.3 mg/kg/dose. For participants > 40 kg, the maximum of dose in the first treatment pair was 12.5 mg per dose. Dose escalation to maximum 0.5 mg/kg/dose was permitted.
  Interventions: Drug: methylphenidate; Other: Placebo
- P-M, P-M, M-P (Experimental): Participants were randomized to receive 3 treatment pairs of placebo (P) then methylphenidate (M) or M then P. Each M or P was given daily for 3 days and therefore treatment duration was 18 days over 3 treatment pairs. M or P was administered orally at a starting dose of 0.3 mg/kg/dose. For participants > 40 kg, the maximum of dose in the first treatment pair was 12.5 mg per dose. Dose escalation to maximum 0.5 mg/kg/dose was permitted.
  Interventions: Drug: methylphenidate; Other: Placebo
- P-M, M-P, M-P (Experimental): Participants were randomized to receive 3 treatment pairs of placebo (P) then methylphenidate (M) or M then P. Each M or P was given daily for 3 days and therefore treatment duration was 18 days over 3 treatment pairs. M or P was administered orally at a starting dose of 0.3 mg/kg/dose. For participants > 40 kg, the maximum of dose in the first treatment pair was 12.5 mg per dose. Dose escalation to maximum 0.5 mg/kg/dose was permitted.
  Interventions: Drug: methylphenidate; Other: Placebo
- M-P, M-P, M-P (Experimental): Participants were randomized to receive 3 treatment pairs of placebo (P) then methylphenidate (M) or M then P. Each M or P was given daily for 3 days and therefore treatment duration was 18 days over 3 treatment pairs. M or P was administered orally at a starting dose of 0.3 mg/kg/dose. For participants > 40 kg, the maximum of dose in the first treatment pair was 12.5 mg per dose. Dose escalation to maximum 0.5 mg/kg/dose was permitted.
  Interventions: Drug: methylphenidate; Other: Placebo
- M-P, P-M, P-M (Experimental): Participants were randomized to receive 3 treatment pairs of placebo (P) then methylphenidate (M) or M then P. Each M or P was given daily for 3 days and therefore treatment duration was 18 days over 3 treatment pairs. M or P was administered orally at a starting dose of 0.3 mg/kg/dose. For participants > 40 kg, the maximum of dose in the first treatment pair was 12.5 mg per dose. Dose escalation to maximum 0.5 mg/kg/dose was permitted.
  Interventions: Drug: methylphenidate; Other: Placebo
- M-P, M-P, P-M (Experimental): Participants were randomized to receive 3 treatment pairs of placebo (P) then methylphenidate (M) or M then P. Each M or P was given daily for 3 days and therefore treatment duration was 18 days over 3 treatment pairs. M or P was administered orally at a starting dose of 0.3 mg/kg/dose. For participants > 40 kg, the maximum of dose in the first treatment pair was 12.5 mg per dose. Dose escalation to maximum 0.5 mg/kg/dose was permitted.
  Interventions: Drug: methylphenidate; Other: Placebo
- P-M, P-M, P-M (Experimental): Participants were randomized to receive 3 treatment pairs of placebo (P) then methylphenidate (M) or M then P. Each M or P was given daily for 3 days and therefore treatment duration was 18 days over 3 treatment pairs. M or P was administered orally at a starting dose of 0.3 mg/kg/dose. For participants > 40 kg, the maximum of dose in the first treatment pair was 12.5 mg per dose. Dose escalation to maximum 0.5 mg/kg/dose was permitted.
  Interventions: Drug: methylphenidate; Other: Placebo
- P-M, M-P, P-M (Experimental): Participants were randomized to receive 3 treatment pairs of placebo (P) then methylphenidate (M) or M then P. Each M or P was given daily for 3 days and therefore treatment duration was 18 days over 3 treatment pairs. M or P was administered orally at a starting dose of 0.3 mg/kg/dose. For participants > 40 kg, the maximum of dose in the first treatment pair was 12.5 mg per dose. Dose escalation to maximum 0.5 mg/kg/dose was permitted.
  Interventions: Drug: methylphenidate; Other: Placebo

INTERVENTIONS:
Drug: methylphenidate
  Other Names: MPH; Ritalin; Methylin; Concerta
Other: Placebo

SUMMARY:
The overall aim of this pilot study is to conduct a combined N-of-1 trial (N-1-T) of MPH (methylphenidate) for amelioration of fatigue in children with cancer, and to evaluate the N-1-T design both for individual clinical decision making and for clinical trials in symptom management in pediatric oncology patients. Because no one knows which of the study options are best, participants will receive liquid MPH on some days and a placebo on other days. We will compare how the participant feels on MPH days with how they feel on placebo days to determine whether MPH makes a difference.

DETAILED DESCRIPTION:
I. To assess the N-1-T as a study design to evaluate a symptom-directed intervention in children with cancer

Primary objective

-To evaluate the feasibility of conducting an N-1-T to evaluate MPH for cancer-related fatigue in children as a group

Secondary objectives

* To evaluate the ability of the N-1-T to assess efficacy of MPH for an individual subject statistically and clinically definite answer (regarding the ability of MPH to reduce fatigue)
* To explore subject/family and oncologist perspectives on N1T participation
* To examine in a preliminary fashion whether there are patient, family, disease or study-related factors that are associated with attrition to help guide future large-scale N1Ts

II. To evaluate MPH for treatment of cancer-related fatigue and related symptoms in children

Primary objective

-To evaluate the effect of MPH on cancer-related fatigue in children based on various assessments including pedsFACIT-F and a unidimensional single-item Likert scale for measuring fatigue

Secondary objective

-To assess the side effect profile of MPH for fatigue in children with cancer

III. To evaluate fatigue assessment tools Primary objective

-To evaluate correlation between fatigue scores

ELIGIBILITY:
Inclusion Criteria:

* Participants must be receiving cancer-directed treatment at Dana-Farber Cancer Institute/Children's Hospital Boston or have advanced cancer
* 7-21 years old
* Laboratory values as outlined in the protocol
* Negative pregnancy test (for females of childbearing potential only)
* Child and at least one parent/legal guardian has spoken and written knowledge of English
* Participant has approximately age-appropriate knowledge of English and is able to understand and complete the single-item Likert scale for rating fatigue
* Baseline pedsFACIT-F score of 20 or greater
* Able to reliably take a liquid enterally
* Physical examination including measurement of pulse and blood pressure conducted within the past 14 days
* If the child is on an opioid analgesic, the primary oncologist does not anticipate a need to increase opioid during the study
* Opioid dose stable for at least 5 days immediately prior to enrollment
* No initiation of or change in the dose of benzodiazepine or other sedative/hypnotic drug in the week prior to enrollment and no forseeable initiation or change during the study
* If currently on an SSRI, SNRI, or tricyclic antidepressant, on a stable dose of the past week
* Participant has telephone access for communication with the study team regarding potential dose adjustments and can provide telephone number and alterative phone number

Exclusion Criteria:

* Participant is regarded by primary oncologist to be at a high likelihood of death within 30 days
* Diagnosis of brain tumor, metastatic disease to the brain, or current active CNS leukemia
* Known history of glaucoma
* Receiving palliative sedation
* Receipt of MPH or any other psychostimulant, alpha-adrenergic medications, neuroleptics, lithium, monoamine oxidase inhibitors, procarbazine or coumadin in the 14 days prior to enrollment
* Significant GI disturbance that would impair absorption of the drug
* History of alcohol or substance abuse in the subject. Subjects living with a household member with a history of alcohol or substance abuse may be excluded if the investigator feels there is a risk of the study medication being abused or diverted
* Documented history of psychotic or bipolar disorder, delirium, major depression, suicidal ideation, aggressive behavior necessitating psychiatric care, or any other psychiatric condition requiring urgent psychiatric evaluation or immediate initiation of pharmacotherapy
* History of tics or Tourette's syndrome
* Prior history of adverse reaction to MPH
* Uncontrolled hypertension
* Cardiomyopathy, serious structural cardiac abnormalities, or history of any of the following: ventricular arrhythmia, myocardial infarction, rheumatic fever, spontaneous or unexplained syncope, exercise-induced syncope, or exercise-induced chest pain.
* Family history of ventricular arrhythmia, a sudden or unexplained event requiring resuscitation or sudden death under age 30 years, known cardiac arrhythmia, hypertrophic cardiomyopathy, or dilated cardiomyopathy.
* Concurrent participation in a study that prohibits enrollment on any other trials involving cancer-directed or symptom-directed therapies, without approval from the study PI
* Prior or current medical condition that, in the opinion of the PI, could be exacerbated by MPH
* Pregnant or breastfeeding women
* HIV-positive individuals on combination antiretroviral therapy
* Treatment of fatigue medications or herbal supplements for fatigue during the 14 days prior to enrollment

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Ullrich, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute/Children's Hospital Boston
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 participants were enrolled between July 2011 and January 2012. Only the arms of these participants are presented.
Period: Overall Study
Arm/Group | M-P, P-M, M-P | P-M, P-M, M-P | P-M, M-P, M-P
Started | 1 | 1 | 1
Evaluable for pedsFACIT-F Score Change | 0 | 1 | 0
Completed | 0 | 1 | 0
Not Completed | 1 | 0 | 1
Not completed — Side Effects | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all enrolled patients.
Groups:
- All Participants: Participants were randomized to receive 3 treatment pairs of placebo (P) then methylphenidate (M) or M then P. Each M or P was given daily for 3 days and therefore treatment duration was 18 days over 3 treatment pairs. M or P was administered orally at a starting dose of 0.3 mg/kg/dose. For participants > 40 kg, the maximum of dose in the first treatment pair was 12.5 mg per dose. Dose escalation to maximum 0.5 mg/kg/dose was permitted.
Arm/Group | All Participants
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 16 [11 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Completion Rate of Two Treatment Pairs Using the N-1-T Design
Description: The feasibility of conducting an N-1-T to evaluate MPH for cancer-related fatigue will be determined by the completion rate of two MPH-placebo pairs.
Time Frame: 18 days
Population: The analysis dataset is comprised of all enrolled patients. Based on the definition of the outcome being evaluated, aggregation of data for all participants is appropriate.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 3
participants | 1

2. Secondary Outcome: Rate of Receiving Clinically Definite Answer Regarding the Ability of Experimental Treatment to Reduce Fatigue Using the N-1-T Design
Description: Efficacy of the N-1-T design is defined as patient providing a clinically definite answer regarding the ability of MPH to reduce fatigue.Based on the definition of the outcome being evaluated, aggregation of data for all participants is appropriate.
Time Frame: 18 days
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Number; unit: participants
Arm/Group | M-P, P-M, M-P | P-M, P-M, M-P | P-M, M-P, M-P
Number analyzed (Participants) | 1 | 1 | 1
participants | 0 | 1 | 0

3. Secondary Outcome: Change Over Treatment Pairs in pedsFACIT-F Score
Description: The pediatric Functional Assessment of Chronic Illness Therapy-Fatigue (pedsFACIT-F) is an 11-item instrument derived from a comprehensive pediatric item bank that assesses fatigue. (Lai et al. Pediatr Hematol Oncol 2007) Measuring fatigue over the past 7 days in a population of pediatric cancer patients, the pedsFACIT-F instrument has a score ranging from 0-44, with a higher score meaning more fatigue. A minimally important difference (MID) was established as 4.7 points.
Time Frame: The pedsFACIT-Fwas administered at baseline and at the end of each treatment pair (TP) and related change in score was calculated for each period: baseline to end of TP 1 (day 6); end of TP 1 to end of TP 2 (day 12); end of TP 2 to end of TP 3 (day 18).
Population: The analysis dataset is comprised of all enrolled patients with data at baseline and end of all treatment pairs.
Measure: Number; unit: units on a scale
Arm/Group | P-M, P-M, M-P
Number analyzed (Participants) | 1
units on a scale
  Change from Baseline to end of Treatment Pair 1 | 4
  Change from end of Treatment Pair 1 to Pair 2 | 2
  Change from end of Treatment Pair 2 to Pair 3 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected continuously during treatment. As noted in limitations, the study did not meet the accrual target due to lack of resources. AE data by individual is not accessible and therefore AE outcomes for the 3 participants are aggregated.
Description: The metabolic/laboratory-other cases were elevated lactate dehydrogenase (LDH), ketonuria and bilirubin in urinalysis. The cardiac-other case was hypertensionsinus tachycardia. The constitutional symptoms-other case was decreased appetite.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=3)
hemoglobin (Blood and lymphatic system disorders) | 1
Mood alteration - anxiety (Psychiatric disorders) | 1
Metabolic/Laboratory-Other (Investigations) | 1
Rigors/chills (General disorders) | 1
Constitutional Symptoms-Other (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
diarrhea (Gastrointestinal disorders) | 2
Creatinine (Investigations) | 1
Alkaline phosphatase (Investigations) | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 2
Neuropathy: cranial - CN VII Motor-face; Sensory-taste (Nervous system disorders) | 1
fatigue (General disorders) | 2
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1
fracture (Injury, poisoning and procedural complications) | 1
Cardiac General-Other (Cardiac disorders) | 1
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2
hypotension (Vascular disorders) | 1
Insomnia (Psychiatric disorders) | 1
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1
PTT (Partial thromboplastin time) (Investigations) | 1
Proteinuria (Renal and urinary disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Infection-Other (Infections and infestations) | 1
Tremor (Nervous system disorders) | 1
Urine color change (Renal and urinary disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to insufficient resources.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No